CLINICAL TRIAL: NCT04599101
Title: Effectiveness of Nasal Suction in Infants With Bronchiolitis Using a NoseFrida vs. Bulb Syringe
Brief Title: Nasal Suction in Infants With Bronchiolitis Using a NoseFrida vs. Bulb Syringe
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to difficulty enrolling
Sponsor: Corewell Health East (Other)
Collaborators: Fridababy (Industry)
Responsible Party: Principal Investigator, Margaret J Menoch, MD, Emergency Medicine Physician, Corewell Health East
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2020-325
Record Dates: First submitted 2020-10-17; First posted 2020-10-22 (Actual); Results first posted 2024-04-04 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Bronchiolitis; Respiratory Disease
Keywords: nasal suction; nasal secretions
MeSH Terms: conditions — Bronchiolitis; Respiration Disorders

STUDY DESIGN:
Intervention Model Description: single site, prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Nasal suction device: Nose Frida (Experimental): Nose Frida nasal suction device to clear nasal secretions
  Interventions: Device: Nose Frida nasal suction device
- Nasal suction device: Bulb (Active Comparator): Bulb syringe suction device to clear nasal secretions
  Interventions: Device: Bulb syringe nasal suction device

INTERVENTIONS:
Device: Nose Frida nasal suction device — Caregivers will be given a Nose Frida device to remove the child's nasal secretions.
  Arms: Nasal suction device: Nose Frida
Device: Bulb syringe nasal suction device — Caregivers will be given a bulb syringe device to remove the child's nasal secretions.
  Arms: Nasal suction device: Bulb

SUMMARY:
This research study will evaluate the difference in effectiveness of nasal suction between two different suction devices (NoseFrida and bulb syringe) in infants that have bronchiolitis. Bronchiolitis (a virus infection that goes into the lungs, which subsequently causes difficulty breathing, difficulty sleeping, and difficulty eating and drinking in children) is a common infection in young children. The caregiver-participants will be supplied with a suction devices (either NoseFrida and bulb syringe suction). The device should be used to clear nasal secretions as needed following discharge from the Emergency Center. The participants will be asked to use either a NoseFrida device or a bulb syringe. Caregivers will monitor how well their baby is breathing, eating/drinking, sleeping and how many times the baby has been seen by a medical provider in the 5 days post discharge from the Emergency Center. Post discharge, caregivers will complete a REDCAP survey asking questions about how their baby has been doing over the first 5 days following hospital discharge. REDCAP survey will be sent day 5 and again on day 7 if not completed. This completes study involvement.

DETAILED DESCRIPTION:
Bronchiolitis is common infection in the small airways of the lungs in the pediatric population. It typically affects children under the age of two years during the fall and winter months.Infants with this condition often have a significant amount of nasal drainage and congestion. Infants are known to be obligate nasal breathers. When the nasal secretions block the nasal airway, then breathing, sleeping, and eating/drinking all become very difficult. For this reason it is very important to have a good method of suctioning out the nose and clearing out the secretions. Historically a baby's nose was suctioned with a bulb syringe. These are still commonly used and are given out in the hospital setting, although there are many other types of devices that have been developed recently that are used for suctioning. One of these devices that has become very common among parents now is called the NoseFrida. It is important to evaluate this device and its efficacy compared to the bulb syringe.

This research study will evaluate the difference in effectiveness of nasal suction between two different suction devices (NoseFrida and bulb syringe) in infants that have bronchiolitis. Bronchiolitis (a virus infection that goes into the lungs, which subsequently causes difficulty breathing, difficulty sleeping, and difficulty eating and drinking in children) is a common infection in young children. Patients will be considered for enrollment in the study based on inclusion/exclusion criteria. The patient's caregiver will be supplied with an information sheet, and any questions will be addressed. Those who verbally consent will be enrolled in the study. After parents or guardians (caregivers) provide informed consent for their child, researchers will review the child's medical record for information regarding their history of respiratory distress. The caregiver will then be supplied with a suction device to be used once they are discharged home. The participants will be asked to use a NoseFrida device or a bulb syringe. The device supplied which is instructed to be used will be dependent on the week of enrollment in the study. Education will be given on how to use their respective the suction device devices. Along with the device, a form (Home monitoring form) will be supplied that will outline what should be monitored while using the device, including: number of days after discharge until respiratory symptoms resolve, number of days until the infant is eating/drinking well, and the number of days until the infant is sleeping well. A REDCAP survey will be emailed to participants after 5 days post discharge and again 7 days post discharge if not completed.

The protocol was revised to supply both nasal suction devices to the participants. However, no data was collected under this revised protocol before termination.

ELIGIBILITY:
Inclusion Criteria:

* Infants 18 months of age or younger
* Evaluated in the Emergency Center at Beaumont, Royal Oak
* Diagnosis of bronchiolitis, or presenting symptoms that are consistent with this diagnosis, such as cough, difficulty in breathing, wheezing, decreased oral intake, Fever
* Initial Emergency Center visit for the current illness

Exclusion Criteria:

* Clinically ill, as defined by: Requiring respiratory support (ex. O2 nasal canula, or HFNC) or Abnormal respiratory rate on most recent measurement, per Pediatric Advanced Life Support (PALS) guidelines: Infant- >53 breaths per minute, Toddler- >37 breaths per minute
* Any history of structural upper airway disease, including Cleft palate, Tracheomalacia/laryngomalacia or Subglottic stenosis
* Previously enrolled in the study

Max Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2020-11-21 (Actual); Primary Completion 2023-04-18 (Actual); Study Completion 2023-04-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margaret J Menoch, Principal Investigator — Beaumont
Locations (1):
- Margaret J Menoch, MD, Royal Oak, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nasal Suction Device: Nose Frida | Nasal Suction Device: Bulb
Started | 12 | 9
Completed | 7 | 4
Not Completed | 5 | 5
Not completed — Lost to Follow-up | 5 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nasal Suction Device: Nose Frida | Nasal Suction Device: Bulb | Total
Number analyzed (Participants) | 12 | 9 | 21
Age, Continuous [Mean (Standard Deviation); unit: months] | 11.3 (2.5) | 8.5 (6.8) | 10.1 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 8
  Male | 7 | 6 | 13
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 12 | 9 | 21

OUTCOME MEASURES:

1. Primary Outcome: Number of Emergency Room Visits
Description: Number of emergency room visits for the same respiratory illness within 5 days following discharge, measured via caregiver response on Redcap survey
Time Frame: 5 days
Population: 5 participants in bulb group and 5 participants in the nose frida group did not complete follow up and no data was collected.
Measure: Number; unit: number of visits
Arm/Group | Nasal Suction Device: Nose Frida | Nasal Suction Device: Bulb
Number analyzed (Participants) | 7 | 4
number of visits | 0 | 0

2. Primary Outcome: Number of Participants Readmitted to Hospital for Respiratory Illness or Dehydration
Description: Number of participants readmitted to Hospital for respiratory illness or dehydration within 5 days following discharge, measured via caregiver response on Redcap survey
Time Frame: 5 days
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nasal Suction Device: Nose Frida | Nasal Suction Device: Bulb
Number analyzed (Participants) | 7 | 4
Participants | 0 | 0

3. Secondary Outcome: Caregiver Device Preference
Description: In response to "Which device did you prefer?" on caregiver survey, caregiver may select NoseFrida, Bulb Syringe, Both, or Neither.
Time Frame: 5 days
Population: This outcome measure was applicable to a protocol revision where participants received both devices. No data was collected under this protocol revision.
Arm/Group | Nasal Suction Device: Nose Frida | Nasal Suction Device: Bulb
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Caregiver Perception of NoseFrida Device Effectiveness
Description: In response to "Which device was more effective in suctioning your baby's nose?" on caregiver survey, responses using a likert scale (0-NoseFrida less effective, 1-NoseFrida equally effective, 2-NoseFrida more effective). A higher score represents higher caregiver perceived effectiveness of NoseFrida
Time Frame: 5 days
Population: as for outcome 3
Arm/Group | Nasal Suction Device: Nose Frida | Nasal Suction Device: Bulb
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Caregiver Perception of Bulb Device Effectiveness
Description: In response to "Which device was more effective in suctioning your baby's nose?" on caregiver survey, responses using a likert scale (0-Bulb Syringe less effective, 1-Bulb Syringe equally effective, 2-Bulb Syringe more effective). A higher score represents higher caregiver perceived effectiveness of bulb syringe
Time Frame: 5 days
Population: as for outcome 3
Arm/Group | Nasal Suction Device: Nose Frida | Nasal Suction Device: Bulb
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Number of Days After Discharge Until Respiratory Symptoms Return to Pre-illness Levels
Description: Number of days after discharge until respiratory symptoms (tachypnea, retractions, increased WOB) return to pre-illness levels.
Time Frame: 7 days
Population: Data was not collected for 9 participants in the bulb group who did not complete follow up. Data was not collected for 9 participants in the nose frida group who did not complete follow up.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Nasal Suction Device: Nose Frida | Nasal Suction Device: Bulb
Number analyzed (Participants) | 3 | 0
days | 1.3 (0.6) |

7. Secondary Outcome: Number of Days After Discharge Until Eating/Drinking Returns to Pre-illness Levels
Description: Number of days after discharge until eating/drinking returns to pre-illness levels
Time Frame: 7 days
Population: No data was collected for 6 participants in the Nose Frida group who did not complete follow up. No data was collected for 5 participants in the Bulb group who did not complete follow up.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Nasal Suction Device: Nose Frida | Nasal Suction Device: Bulb
Number analyzed (Participants) | 6 | 4
days | 1.5 (1.2) | 1.0 (0)

8. Secondary Outcome: Number of Days After Discharge Until Sleeping Returns to Pre-illness Levels
Description: Number of days after discharge until sleeping returns to pre-illness levels
Time Frame: 7 days
Population: No data was collected for 8 participants in the Nose Frida group who did not complete follow up. No data was collected for 6 participants in the Bulb group who did not complete follow.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Nasal Suction Device: Nose Frida | Nasal Suction Device: Bulb
Number analyzed (Participants) | 4 | 3
days | 1.0 (0) | 1.0 (0)

9. Secondary Outcome: Parental Satisfaction on Suction Product Efficacy
Description: Parental satisfaction on a likert scale (1-strongly disagree, 2-disagree, 3-undecided, 4-agree, 5-strongly agree) for the question "Does this product suction babies nose well?"
Time Frame: 7 days
Population: No data collected for 8 participants in the Nose Frida group who did not complete follow up. No data collected for 7 participants in the Bulb group who did not complete follow up.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Nasal Suction Device: Nose Frida | Nasal Suction Device: Bulb
Number analyzed (Participants) | 4 | 2
score on a scale | 4 [3 to 5] | 4.5 [3 to 5]

10. Secondary Outcome: Parental Satisfaction on Ease of Use
Description: Parental satisfaction on a likert scale (1-strongly disagree, 2-disagree, 3-undecided, 4-agree, 5-strongly agree) for the question "Is this product easy to use?"
Time Frame: 7 days
Population: as for outcome 9
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Nasal Suction Device: Nose Frida | Nasal Suction Device: Bulb
Number analyzed (Participants) | 4 | 2
score on a scale | 4.5 [3 to 5] | 4.5 [3 to 5]

11. Secondary Outcome: Participant Recommendation to Other Parents
Description: Parental agreement on a likert scale (1-strongly disagree, 2-disagree, 3-undecided, 4-agree, 5-strongly agree) for the statement "I would recommend this product to other parents."
Time Frame: 7 days
Population: as for outcome 9
Measure: Median (Full Range); unit: score on a scale
Arm/Group | Nasal Suction Device: Nose Frida | Nasal Suction Device: Bulb
Number analyzed (Participants) | 4 | 2
score on a scale | 4.5 [4 to 5] | 4.5 [3 to 5]

ADVERSE EVENTS:
Time Frame: 7 days
Arm/Group | Nasal Suction Device: Nose Frida | Nasal Suction Device: Bulb
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/9
Other Adverse Events (participants affected / at risk) | 0/12 | 0/9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2020-10-07): https://cdn.clinicaltrials.gov/large-docs/01/NCT04599101/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-04): https://cdn.clinicaltrials.gov/large-docs/01/NCT04599101/SAP_001.pdf
  • Informed Consent Form (2023-09-15): https://cdn.clinicaltrials.gov/large-docs/01/NCT04599101/ICF_002.pdf